CLINICAL TRIAL: NCT06855758
Title: Effect of Terlipressin for Intraoperative Blood Pressure Management in Kidney Transplantation, a Double-blind Randomized Controlled Trial
Brief Title: Effect of Terlipressin for Intraoperative Blood Pressure Management in Kidney Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-P2-023-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant; Delayed Graft Function; Intraoperative Hypotension
MeSH Terms: conditions — Delayed Graft Function | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dopamine (No Intervention): Continuous using of dopamine as blood pressure regulation after anesthesia, with dosage adjusted according to intraoperative needs
- terlipressin + dopamine (Experimental): Terlipressin was given before the graft circulation was established while continuous using of dopamine during the whole operation
  Interventions: Drug: terlipressin

INTERVENTIONS:
Drug: terlipressin — Terlipressin was given prior to the opening of the graft circulation (with the possibility of reperfusion hypotension) when the blood pressure is suboptimal and does not respond well to dobutamine or fluid volume resuscitation. 1 mg terlipressin + 100 ml of sodium chloride injections was given for intravenous infusion.
  Arms: terlipressin + dopamine

SUMMARY:
Prospective double blind randomized controlled trial. By randomizing patients undergoing kidney transplantation into a conventional catecholamine drug (dobutamine) blood pressure maintenance group and a terlipressin-complexed dobutamine group, the investigators compared the effect of intraoperative blood pressure maintenance and the dosage of the vasoactive drug, postoperative graft function, delayed graft function, and other related complications between the two groups, in order to demonstrate whether the use of terlipressin for blood pressure regulation during kidney transplantation is superior to the existing treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease aged 18 years or above

Exclusion Criteria:

* simultaneous multiple organ transplantation
* known allergy to study medication
* known pregnancy status
* cancellation of surgery due to grafts or personal reasons
* persistent severe preoperative hypertension that may not require intraoperative supportive therapy with vasoactive medications
* any other reason that the supervising physician or the anesthesiologist on duty think the patient is not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Delayed graft function | within the first 7 days after op
  need kidney replacement in the first 7 days after op

CONTACTS AND LOCATIONS:
Overall Officials: Fushan Xue, Principal Investigator — Department of Anesthesiology, Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Selected statistics related to outcomes
Supporting Information: Study Protocol, SAP
Time Frame: after published
Access Criteria: Investigators who submitting research proposals and signing agreements of data using with corresponding authors